CLINICAL TRIAL: NCT06715878
Title: Zero Ischemia Robot-Assisted Microwave Ablation Assisted Suture-less Enucleation of Renal Cell Carcinoma With T1 Stage: A Randomized Clinical Trial
Brief Title: Zero Ischemia Robot-Assisted MWA Assisted Suture-less Tumor Enucleation of RCC With T1 Stage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIRACLE
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Kidney Neoplasms
Keywords: Microwave ablation; Nephronsparing surgery; Zero ischemia; suture less
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zero Ischemia suture-less group (Experimental): Patients with T1 Stage renal cell carcinoma undergoing Zero Ischemia, Robot-Assisted Microwave Ablation assisted suture-less tumor Enucleation.
  Interventions: Procedure: Zero Ischemia Robot-Assisted Laparoscopic Microwave Ablation Assisted suture-less Enucleation
- robotic-assisted partial nephrectomy group (Active Comparator): Patients with T1 stage Renal Cell Carcinoma undergoing traditional robotic-assisted partial nephrectomy.
  Interventions: Procedure: robotic-assisted laparoscopic partial nephrectomy

INTERVENTIONS:
Procedure: Zero Ischemia Robot-Assisted Laparoscopic Microwave Ablation Assisted suture-less Enucleation — Under the visualization of ultrasound contrast imaging through the operative channel, a microwave ablation probe was inserted into the tumor (at the interface between the tumor and kidney, close to the tumor base). The microwave ablation device was used, with a power setting of 70 W for initiating microwave ablation. Depending on the tumor volume and depth, 1-3 ablation cycles were performed, with each cycle lasting 1-3 minutes. After reaching the pseudocapsule of the tumor, a combination of blunt dissection, sharp cutting, and blunt dissection was employed to separate the tumor from the renal parenchyma . The renal artery was not occluded during the procedure.If intraoperative injury to the collecting system is suspected, the collecting system should be sutured normally, while simultaneously suturing the outer layer of renal parenchyma to prevent urine leakage.
  Arms: Zero Ischemia suture-less group
Procedure: robotic-assisted laparoscopic partial nephrectomy — robotic-assisted laparoscopic partial nephrectomy
  Arms: robotic-assisted partial nephrectomy group

SUMMARY:
Zero ischemia laparoscopic radio frequency ablation assisted tumor enucleation has been proved to enable tumor excision with relatively better renal function preservation comparing with conventional laparoscopic partial nephrectomy for T1a renal cell carcinoma (RCC) in a randomized clinical trial in single center. The investigators want to explore this technique to robotic surgery and add suture-less technique to T1 RCC patients in randomized clinical trial.

DETAILED DESCRIPTION:
Zero ischemia laparoscopic radio frequency ablation assisted tumor enucleation has been proved to enable tumor excision with relatively better renal function preservation comparing with conventional laparoscopic partial nephrectomy for T1a renal cell carcinoma (RCC) in a randomized clinical trial in single center. The investigators want to explore this technique to robotic surgery and add suture-less technique to T1 RCC patients in randomized clinical trial. This project is based on the previous research and aims to develop an approach of the combination of intraoperative real time contrast-enhanced ultrasonography technology, sutureless technology and the zero ischemia robot-Assisted tumor enucleation of the kidney. By using the real time contrast-enhanced ultrasonography technology, the current shortcomings of the zero ischemia laparoscopic radio frequency ablation assisted tumor enucleation were overcome. The degree of elimination was monitored during surgery to avoid excessive bleeding caused by insufficient ablation during the surgery. Beside, the difficulty of zero ischemia laparoscopic radio frequency ablation is reduced, and doctors can quickly grasp the learning curve of this technology.

ELIGIBILITY:
Inclusion Criteria:

1. patients with sporadic, unilateral, newly diagnosed T1 presumed renal cell carcinoma
2. patients scheduled for robot-assisted laparoscopic nephron sparing surgery
3. patients with normal contralateral renal function (differential renal function of >40% as determined by radionuclide scintigraphy)
4. patients agreeable to participate in this long-term follow-up study

Exclusion Criteria:

1. patients' age >80 years
2. patients with other renal diseases (including kidney stone, glomerular nephritis, etc.)which might affect the renal function of the operative kidney
3. patients not able to tolerate the robot-assisted laparoscopic procedure
4. patients with previous renal surgery or history of any inflammatory conditions of the operative kidney
5. patients with the renal tumor involving urinary collecting system or distance from the tumor edge to the collecting system ≤ 4 mm

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The absolute change in glomerular filtration rate (GFR) of the affected kidney | baseline and 12 months
  12 months minus baseline
The changes of estimated GFR (eGFR) | baseline and 12 months
  12 months minus baseline

SECONDARY OUTCOMES:
estimated blood loss | during surgery
changes in GFR of total kidneys by renal scintigraphyby | baseline and 12 months
surgical margin | postoperative up to 2 weeks after surgery
postoperative complications | postoperative up to 30 days
progression-free survival | 12 months
local recurrence | 12 months
operative time | During surgery
Hospital stay time | The time from the surgery day to patient discharge, up to 2 weeks
changes in GFR of total kidneys by renal scintigraphyby of 3 month | baseline and 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics Committee of Shanghai Renji Hospital, Shanghai, China